CLINICAL TRIAL: NCT06126887
Title: Evaluation of Efficacy and Comfort: A Randomized Clinical Trial on the Incrediwear Back Brace in Patients With Chronic Lower Back Pain
Brief Title: Evaluation of Efficacy and Comfort: A Trial on the Incrediwear Back Brace in Patients With Chronic Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00391930
Record Dates: First submitted 2023-10-29; First posted 2023-11-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain; Back Pain
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Incrediwear Daytime (Experimental): Incrediwear back brace worn 7AM-7PM (against skin)
  Interventions: Device: Incrediwear Daytime Back Brace
- Incrediwear Sham Daytime (Sham Comparator): Incrediwear sham back brace worn 7AM-7PM (against skin)
  Interventions: Device: Incrediwear Sham Daytime Back Brace
- Control Daytime (Placebo Comparator): Standard-issue brace (e.g. Horizon Lumbar Brace (Aspen Medical Products, LLC)) worn 7AM-7PM
  Interventions: Device: Control Daytime Back Brace
- Incrediwear 24 hour (Active Comparator): Incrediwear back brace worn 7AM-7PM (against skin). Incrediwear waist sleeve worn 7PM-7AM (against skin)
  Interventions: Device: Incrediwear 24 Hour Back Brace

INTERVENTIONS:
Device: Incrediwear Daytime Back Brace — Incrediwear Daytime Back Brace
  Arms: Incrediwear Daytime
Device: Incrediwear Sham Daytime Back Brace — Incrediwear Sham Daytime Back Brace
  Arms: Incrediwear Sham Daytime
Device: Control Daytime Back Brace — Control Daytime Back Brace
  Arms: Control Daytime
Device: Incrediwear 24 Hour Back Brace — Incrediwear 24 Hour Back Brace
  Arms: Incrediwear 24 hour

SUMMARY:
The investigators hypothesize that the utilization of Incrediwear's Back Brace, compared to a sham brace and a standard-issue brace, will lead to better brace adherence, increased patient satisfaction, reduced pain medication usage, and improved functional disability among non-surgical chronic LBP patients.

DETAILED DESCRIPTION:
Problem: Chronic low back pain (LBP) affects a substantial portion of the population and often leads to decreased functional ability and increased pain medication usage. While back braces have been recommended as part of LBP management, their efficacy and impact on patient outcomes remain uncertain.

Research Hypothesis: The investigators hypothesize that the utilization of Incrediwear's Back Brace, compared to a sham brace and a standard-issue brace, will lead to better brace adherence, increased patient satisfaction, reduced pain medication usage, and improved functional disability among non-surgical chronic LBP patients.

Importance of the Research: This randomized clinical trial aims to assess the efficacy of Incrediwear's Back Brace in improving patient outcomes for chronic LBP. The study will provide valuable insights into the utilization patterns and adherence of back braces, patient satisfaction with treatment protocols, and the impact of brace usage on pain medication consumption and functional disability. By evaluating these factors through a controlled trial, the investigators seek to enhance the understanding of effective LBP management strategies, potentially reducing the burden of chronic LBP on patients and healthcare systems.

The study will be conducted under the guidance of Dr. Akhil Chhatre, Principal Investigator at the Department of Physical Medicine and Rehabilitation, Johns Hopkins University School of Medicine. The research will involve 100 non-surgical chronic LBP patients meeting specific inclusion criteria. The patients will be randomly assigned to one of four study groups, and data will be collected through phone calls over a full 4-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age > 18
* Has undergone treatment for an initial episode of nonspecific low back pain (LBP) lasting > 1 month, with one of the following causative "Principle Diagnoses":
* Disc herniation
* Facet arthropathy
* Compression fracture
* Spondylolisthesis
* Sacroiliac joint dysfunction
* Scoliosis
* Mild to moderate central spinal stenosis
* Lumbar spondylosis
* Degenerative changes, not otherwise specified
* Utilize pain medication (including Step I or II analgesics, NSAIDs, Benzodiazepines) at least weekly for their LBP
* Subject report a VAS pain score at the time of consent greater than three (>3) out of ten (10)
* Recommended a back brace for LBP management
* Provide written consent for participation
* Subject available for phone calls after 6PM

Exclusion Criteria:

* Severe central spinal stenosis
* Focal lower extremity weakness
* LBP radiating beyond the knee and/or accompanied by neurological signs (including sciatica)
* Spinal operation within 5 years preceding the study date
* Secondary LBP due to a work accident (e.g. workers comp)
* History of spinal arthrodesis
* LBP with an inflammatory, tumor, or infectious cause
* Contraindications to: Step I or II analgesics, NSAIDs, Benzodiazepines
* Diagnosed peripheral arterial disease
* Diabetes
* Higher functions do not enable proper comprehension of protocol or reliable data recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
User Evaluation of Satisfaction as assessed by the Quebec User Evaluation of Satisfaction with Assistive Technology 2.0 (QUEST 2.0) | 1 month
  Satisfaction (Quebec User Evaluation of Satisfaction with Assistive Technology 2.0 [QUEST 2.0] score). The score ranges from 1-5 with 1 being not satisfied at all to 5 being very satisfied
Brace and sleeve utilization | 1 month
  Self-reported hours worn
Pain medication name | 1 month
  The investigators aim to explore the effects of brace utilization on pain medication use. The investigators will document the pain medication name
Functional disability status as assessed by the Oswestry Disability Index (ODI) | 1 month
  Oswestry Disability Index (ODI). A total score of 0-4 (no disability), 5-14 (mild disability), 15-24 (moderate disability), 25-34 (severe disability), 35-50 (completely disabled)
Pain as assessed by the Visual Analogue Scale (VAS) | 1 month
  Visual Analogue Scale (VAS) and frequency (ordinal scale). 0 = no pain and 10 = pain as bad as it could possibly be
Pain medication dosage used | 1 month
  The investigators aim to explore the effects of brace utilization on pain medication use. The investigators will document the pain medication dosage used

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Chhatre, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Health Care & Surgery Center - Howard County Medical Center, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided